CLINICAL TRIAL: NCT01098942
Title: Effects of Bariatric Surgery on Skeletal Health
Brief Title: Bariatric Surgery and Skeletal Health
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elaine W. Yu, Co-investigator, Massachusetts General Hospital
Other Study IDs: 2009P001445
Record Dates: First submitted 2010-04-02; First posted 2010-04-05 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Morbid Obesity
Keywords: bariatric surgery
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgical: Roux-en-Y gastric bypass surgery
- Non-surgical: Non-surgical lifestyle weight management

SUMMARY:
Bone loss may occur after bariatric (weight loss) surgery, but standard methods of measuring bone density in obese patients are potentially inaccurate. This study uses quantitative computed tomography to examine changes in bone mineral density after bariatric surgery. We are also studying mechanisms which may explain bone loss after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Either scheduled for Roux-en-Y Gastric Bypass surgery or enrolled in a lifestyle weight management program

Exclusion Criteria:

* Weight ≥ than 450 lbs
* Postmenopausal women
* Significant heart, kidney, liver, or malignant disease
* Current disorders known to affect bone
* Use of medications known to affect bone for more than 7 days in the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese adults
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-08 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Changes in bone mineral density by dual-energy x-ray absorptiometry (DXA) and quantitative computed tomography (QCT) | 1 year

SECONDARY OUTCOMES:
Changes in serum and/or urine indices of bone formation and bone resorption, such as aminoterminal propeptide of type I collagen [PINP], osteocalcin, C-telopeptide cross-links [CTX]) | 1 year
Changes in bone microarchitecture by high-resolution peripheral quantitative computed tomography (HR-pQCT) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joel S. Finkelstein, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - MGH, Boston, Massachusetts

REFERENCES:
- [Derived] Yu EW, Bouxsein ML, Putman MS, Monis EL, Roy AE, Pratt JS, Butsch WS, Finkelstein JS. Two-year changes in bone density after Roux-en-Y gastric bypass surgery. J Clin Endocrinol Metab. 2015 Apr;100(4):1452-9. doi: 10.1210/jc.2014-4341. Epub 2015 Feb 3. PMID 25646793
- [Derived] Yu EW, Bouxsein ML, Roy AE, Baldwin C, Cange A, Neer RM, Kaplan LM, Finkelstein JS. Bone loss after bariatric surgery: discordant results between DXA and QCT bone density. J Bone Miner Res. 2014 Mar;29(3):542-50. doi: 10.1002/jbmr.2063. PMID 23929784